CLINICAL TRIAL: NCT05768620
Title: Active Navigation Training: an Innovative Embodied-based Training System for Spatial Navigation in Aging
Brief Title: Active Navigation Training
Acronym: ANTaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 39M801
Record Dates: First submitted 2023-02-22; First posted 2023-03-14 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Mild Cognitive Impairment; Spatial Navigation
Keywords: virtual reality
MeSH Terms: conditions — Cognitive Dysfunction; Spatial Navigation | interventions — Caves

STUDY DESIGN:
Intervention Model Description: Proof-of-concept trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAVE (Experimental): 10 immersive virtual reality sessions to train spatial memory
  Interventions: Other: CAVE
- TAU (Active Comparator): 10 paper and pencil sessions to train spatial memory
  Interventions: Other: TAU

INTERVENTIONS:
Other: CAVE — The training is designed to train spatial navigation and memory and in particular egocentric and allocentric processes
  Arms: CAVE
Other: TAU — This is the usual care used to train visuospatial processes
  Arms: TAU

SUMMARY:
Pilot testing and development of an immersive virtual reality system for spatial navigation training in mild cognitive impairment syndrome.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of mild cognitive impairment
* absence of severe cognitive deterioration as assessed by the Italian version of the MMSE (Magni et al. 1996)
* age ≥ 60

Exclusion Criteria:

* the presence of acute stroke/transient ischemic attack;
* the presence of other concomitants severe neurological/psychiatric diseases;
* history of traumatic brain injury with loss of consciousness;
* physical/functional deficits that could affect the use of immersive virtual reality;
* severe visual deficiency;
* the presence of recurrent vertigo.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Corsi supra-span test | After 10 training sessions (3/4 weeks approx.) and after 3-month follow-up
  Scores range from 0 to 29.16, higher scores indicate better visuospatial learning
Change in Manikin Test | After 10 training sessions (3/4 weeks approx.) and after 3-month follow-up
  Scores range from 0 to 1, higher scores indicate better visuospatial mental rotation

SECONDARY OUTCOMES:
Trail-making test part A and B | After 10 training sessions (3/4 weeks approx.) and after 3-month follow-up
Raccontino (6 Dicembre) (immediate-delayed-forgetting) | After 10 training sessions (3/4 weeks approx.) and after 3-month follow-up
Mini-mental state examination | After 10 training sessions (3/4 weeks approx.) and after 3-month follow-up
Digit span forward | After 10 training sessions (3/4 weeks approx.) and after 3-month follow-up
Corsi Block Tapping | After 10 training sessions (3/4 weeks approx.) and after 3-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Cosimo Tuena, Milan, Lombardy, Italy